CLINICAL TRIAL: NCT04131283
Title: Evidence of Spreading Vasoconstriction in Human Gingiva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Vag Janos, Principal Investigator, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1/2019
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Vasoconstriction; Oral Soft Tissue Conditions; Dental and Gingival Conditions
Keywords: spreading vasoconstriction; gingival microcirculation
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epinephrine effect throught keratinized ginigva (Experimental): 1 mg/ml epniephrine vs physiologocal saline
  Interventions: Drug: Epinephrine
- Epinephrine effect throught gingival sulcular epithelium (Experimental): 1 mg/ml epniephrine vs physiologocal saline
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Epinephrine — Vasoconstrictor solution is applied on the surface of the attached gingiva and on the gingival sulcus.
  Other Names: retrograde vasoconstriction

SUMMARY:
The aim of this study is to observe the mechanism of spreading vasoconstriction in human healthy gingiva. Epinephrine solution is applied on the attached gingiva in group "A" and on the surface of the tooth next to the ginvial sulcus in group "B". The different placement of the solution causes different effect in the microcirculation.

DETAILED DESCRIPTION:
Spatial regulation of gingival microcirculation has not been revealed yet. Although this could be an important mechanism to protect gingiva as it is exposed to mechanical, chemical, thermal etc. irritation during whole life. It is especially important during flap surgery. Laser Speckle Contrast Imaging (LSCI) is novel non-invasive method with high spatio-temporal resolution, therefore it allows us to study remote effect of local vasoconstriction such as spreading vasoconstriction in human gingiva.

The epinephrine is a daily used vasoconstrictor material in dentistry and it will be used to trigger remote effect on gingiva. Epinephrine in 1 mg/ml concentration. Solution will be dropped on the gingiva at tooth 12 in a fabricated leakage proof well attached to 2mm above the marginal gingiva in group "A". The solution will be dropped on the surface of tooth 12 next to the sulcus into the well in case of group "B". The changes of the blood flow will be monitor at the test side with surrounding gingival area by LSCI. The control side in each case will be - appropriately to the test side - at tooth 21 with phisiologocal saline.

ELIGIBILITY:
Inclusion Criteria:

* at least 5 mm keratinized gingiva at the upper front teeth
* general health

Exclusion Criteria:

* pregnancy, breast-feeding
* any medication
* smoking, gingivitis, caries and coronal restoration with insufficient marginal integrity

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Blood flow change after application of epinephrine | 30 minutes
  The change in blood flow will be measured after locally applied epinephrine at the site fo application and at the remote sites

SECONDARY OUTCOMES:
Comparsion of the change in blood flow between genders | 30 minutes
  The maximal blood flow changed assessed in primary outcome will be split into two groups based on gender. The change will be compared between males and females.

OTHER OUTCOMES:
Correlation between the change in blood flow and gingival thickness | 5 minutes
  The biotpye will be assessed by measurement of gingival thickness by an ultrasonic devices. The correlation between thickness and maximal vasodilation will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Janos Vag, Budapest, Hungary

REFERENCES:
- [Derived] Vag J, Ganti B, Mikecs B, Szabo E, Molnar B, Lohinai Z. Epinephrine penetrates through gingival sulcus unlike keratinized gingiva and evokes remote vasoconstriction in human. BMC Oral Health. 2020 Nov 4;20(1):305. doi: 10.1186/s12903-020-01296-z. PMID 33148235